CLINICAL TRIAL: NCT05859191
Title: Study of Neonatal Immunoglobulin G (IgG) Fc Receptor (FcRn) Expression in Natural Killer T Cells Expressing an Invariant T Receptor (iNKT): Implication in the Pathophysiology of Systemic Lupus
Brief Title: Study of Neonatal IgG Fc Receptor Expression in Natural Killer T Cells Expressing an Invariant T Receptor : Implication in the Pathophysiology of Systemic Lupus
Acronym: FiNKLUPUS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Tours (Other)
Collaborators: Research Center for Respiratory Diseases, Inserm U1100 (Unknown)
Responsible Party: Sponsor
Other Study IDs: DR230103-FiNK LUPUS
Record Dates: First submitted 2023-05-03; First posted 2023-05-15 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-09

CONDITIONS: Systemic Lupus Erythematosus; Physiopathology
Keywords: lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Three extra tubes of blood will be taken at each consultation or inpatient visit when routine blood samples are taken as part of lupus monitoring.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LUPUS PATIENTS: Three extra tubes of blood will be taken at each consultation or inpatient visit when routine blood samples are taken as part of lupus monitoring.
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — Three extra tubes of blood will be taken at each consultation or inpatient visit when routine blood samples are taken as part of lupus monitoring.

SUMMARY:
This study evaluates the variation of expression of the neonatal Fc receptor (FcRn) in Natural Killer T Cells Expressing an Invariant T Receptor (iNKT) and monocytes along with the surface expression of Fc gamma type II receptor (RII) and RIII in active or newly diagnosed lupus patients compared to inactive lupus patients.

DETAILED DESCRIPTION:
The role of FcRn in autoimmune diseases remains to be clarified, but it has been implicated in numerous pathophysiological mechanisms, notably in the management of immune complexes or the recycling of autoantibodies. In humans, this role in the metabolism of autoantibodies has recently led to the development of therapeutic antibodies for autoimmune diseases such as autoimmune thrombocytopenia and myasthenia.

The lupus erythematosus is an auto-immune disease mediated by IgG and immune complexes characterized by a high diversity of autoantibodies and a large dysregulation of the immune system in all it's components, one of them being iNKT cells.

Studies in patients or in lupus mouse models have shown a decrease in iNKT cells correlated with disease activity as well as tissue infiltration in relation to clinical manifestations. Their actual role in this pathology remains to be clarified between regulatory or pro-inflammatory effect.

The possible role of iNKT as a regulatory cell in lupus pathology and the possible involvement of FcRn in their development reinforces the interest of their simultaneous study in humans.

The aim of this study will be to evaluate the impact of the expression of FcRn and other Fc gamma receptors cooperating with FcRn (Fc gamma RII and RIII) in iNKT cells in lupus patients in relation to disease activity and therapy. This study will be conducted in parallel on monocytes, cells involved in the metabolism of immune complexes and likely to be activated by iNKT cells. These results will be compared to healthy controls and integrated into mechanistic studies in a mouse model.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of definite systemic lupus which may be associated with secondary antiphospholipid syndrome and/or secondary Gougerot-Sjögren's
* Lupus patient, newly diagnosed or known, untreated or in relapse
* Lupus patient considered stable by the treating practitioner
* Requiring blood sampling for follow-up

Exclusion Criteria:

* Main autoimmune disease other than lupus
* Patient under legal protection, guardianship or curators
* Opposition to data processing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with systemic lupus
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-07-21 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
FcRn Expression analysis in Circulating iNKT lymphocytes | through study completion, an average of 3 year
  by flow cytometry (mean fluorescence intensity)
FcRn Expression analysis in circulating monocytes | through study completion, an average of 3 year
  by flow cytometry (mean fluorescence intensity)
FcgammaRII Expression analysis in Circulating iNKT lymphocytes | through study completion, an average of 3 year
  by flow cytometry (mean fluorescence intensity)
FcgammaRII Expression analysis in circulating monocytes | through study completion, an average of 3 year
  by flow cytometry (mean fluorescence intensity)
FcgammaRIII Expression analysis in Circulating iNKT lymphocytes | through study completion, an average of 3 year
  by flow cytometry (mean fluorescence intensity)
FcgammaRIII Expression analysis in in circulating monocytes | through study completion, an average of 3 year
  by flow cytometry (mean fluorescence intensity)

SECONDARY OUTCOMES:
corticotherapy | through study completion, an average of 3 year
  data collected from patient medical file
hydroxychloroquine | through study completion, an average of 3 year
  data collected from patient medical file
immunosuppressants outside of biotherapy: methotrexate, azathioprine, mycophenolate mofetil | through study completion, an average of 3 year
  data collected from patient medical file
biotherapy: belimumab and rituximab | through study completion, an average of 3 year
  data collected from patient medical file
lupus disease activity | through study completion, an average of 3 year
  assessed with the Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K). The score ranging from 0 (no activity) to 105
albumin and IgG levels | through study completion, an average of 3 year
  by immunonephelometry

CONTACTS AND LOCATIONS:
Overall Officials: Yanis RAMDANI, Principal Investigator — CHRU de Tours
Locations (1):
- University Hospital, Tours, France

IPD SHARING:
Plan to Share IPD: Undecided